CLINICAL TRIAL: NCT00570648
Title: A Prospective Study of the Effect of Topical Sodium Hyaluronate Immediately Post-PKP on Time to Reepithelialization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Christopher Ketcherside, MD, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13114
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-08

CONDITIONS: Corneal Transplantation
Keywords: Corneal transplantation
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 1% sodium hyaluronate (Healoon) applied at the end of surgery to the surface of the corneal transplant
  Interventions: Drug: sodium hyaluronate
- 2 (No Intervention): Nothing applied at the end of surgery

INTERVENTIONS:
Drug: sodium hyaluronate — 1% sodium hyaluronate applied at the end of corneal transplant surgery. The amount will be determined on how much is necessary to cover the ocular surface.
  Other Names: Healon
  Arms: 1

SUMMARY:
Hypothesis: 1% sodium hyaluronate (Healon), applied at end of surgery to the surface of a corneal transplant will not shorten graft reepithelialization time when compared to coating with nothing. We also wish to measure and compare visual acuity in this immediate post operative period. We also wish to assess the safety of using this agent on the epithelium post-operatively.

We will recruit 50 high risk patients (see inclusion criteria) here at the University of Virginia to randomly receive nothing or sodium hyaluronate (Healon) on the ocular surface at the end of surgery, and follow time to reepithelialization of the corneal transplant grafts.

DETAILED DESCRIPTION:
Corneal transplant is one of the most common transplant procedures, with over 32,000 recipients in the United States in 2005 and a similar number estimated in 2006. The immediate post-operative period is very important in determining the quality of the graft and often its overall chance of survival. The corneal epithelium is replaced by the recipient epithelium after transplant and this should usually take place in no more than 1 week. This reepithelialization is very important for healing, recovery of the epithelial barrier against infectious agents, and for recovery of vision through the graft. Grafts that take longer to heal can invite not only infection and hinder visual recovery, but be permanently scarred, thinned, and even perforate/fail. Thus rapid reepithelialization is crucial. This becomes even more crucial for monocular patients who need quick recovery.

Currently there is no universal agent that is used to coat the surface at the end of surgery before patching. Previous animal studies have shown that sodium hyaluronate will promote rapid migration of cells as well as stimulate cell proliferation leading to rapid wound closure (1,2). In 1987 one smaller study showed that topical sodium hyaluronate (Healon) may foster improved epithelial healing but it was used intraoperatively and presented technical challenges (3). A more recent non-randomized, retrospective study found that sodium hyaluronate at the end of surgery to coat the ocular surface shortened reepithelialization time. This was in comparison to dexamethasone/oxytetracycline ointment and neomycin/dexamethasone drops, both of which hinder reepithelialization (4). To date we know of no prospective, randomized, double-blinded studies that compare the application of sodium hyaluronate versus nothing (currently the practice at UVA).

ELIGIBILITY:
Inclusion Criteria:

* The patients considered for enrollment must be scheduled for penetrating keratoplasty.
* Any high risk patient requiring penetrating keratoplasty.

Criteria for high risk include one of the following:

* Prior failed corneal graft in the operative eye
* Being treated for dry eye at time of surgery
* Having 2 or more quadrants of corneal vascularization
* Having another procedure performed on same eye at time of PKP

Exclusion Criteria:

* Does not meet one of the criteria for high risk
* Known hypersensitivity to hyaluronate preparations
* Allergic to avian proteins, feathers, or egg products
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-06; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Time to graft reepithelialization | weekly until total reepithelialization occurs

SECONDARY OUTCOMES:
Visual acuity | 24 hours post-op and weekly until reepithelialization occurs
safety | 24 hours then weekly until reepithelialization occurs

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ketcherside, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States